CLINICAL TRIAL: NCT07031570
Title: Retrospective Evaluation of the Efficacy and Safety of Drug-Eluting Bead Transarterial Chemoembolization (DEB-TACE) Combined With Hepatic Arterial Infusion Chemotherapy (HAIC) Versus HAIC Alone in Patients With Unresectable Colorectal Cancer Liver Metastases
Brief Title: Efficacy and Safety of DEB-TACE Combined With HAIC Versus HAIC Alone in Patients With Unresectable CRLM
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zhu Xu, Director , Dept of Interventional Therapy, Peking University Cancer Hospital & Institute
Other Study IDs: CRLM-DEBTACE-HAIC
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Metastatic
Keywords: CRLM; DEB-TACE; HAIC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observed group: the patient treated with DEB-TACE combined with HAIC
- Control group: the patient treated with HAIC only

SUMMARY:
Retrospective evaluation of the efficacy and safety of DEB-TACE combined with HAIC versus HAIC alone in patients with unresectable colorectal liver metastases (CRLM)

DETAILED DESCRIPTION:
This study is a retrospective, non-randomized, single-arm, single-center clinical study. Patients who received DEB-TACE combined with HAIC or HAIC alone were screened from the treatment records of the Department of Interventional Radiology at Peking University Cancer Hospital between March 2015 and December 2023. The study aims to observe treatment efficacy, disease progression, and postoperative adverse reactions to evaluate the effectiveness and safety of combination therapy versus HAIC alone in patients with colorectal liver metastases (CRLM). Analyses will be conducted based on various parameters, including but not limited to HAIC perfusion regimens and drug-eluting bead tumor characteristics.

The primary endpoint of the study is progression-free survival (PFS). Secondary endpoints include overall survival (OS), objective response rate (ORR), disease control rate (DCR), and safety. PFS is defined as the time from the first DEB-TACE plus HAIC or HAIC-alone treatment to disease progression. PFS will be categorized into intrahepatic PFS and overall PFS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. No gender restriction
3. Pathologically or clinically diagnosed with colorectal liver metastases
4. Imaging data available within 31 days prior to enrollment, with at least one measurable lesion (according to RECIST criteria)
5. Patients received only DEB-TACE combined with HAIC or HAIC alone during the observation period
6. Child-Pugh classification A or B
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

1. Presence of treatment risks or contraindications to DEB-TACE combined with HAIC or HAIC alone.
2. Concurrent diagnosis of other malignancies.
3. Underwent other local treatment modalities during the observation period.
4. DEB-TACE combined with HAIC or HAIC alone was used as postoperative adjuvant therapy.
5. Missing relevant examination results before or after treatment.
6. Incomplete imaging data, making response evaluation impossible.
7. Follow-up failure due to incorrect or missing patient information, loss to follow-up, or patient refusal.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal liver metastases who received DEB-TACE combined with HAIC or HAIC alone at the Department of Interventional Radiology, Peking University Cancer Hospital, between March 2015 and December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy-PFS | 6-8 weeks after each treatment
  PFS is defined as the time from the date of the first DEB-TACE combined with HAIC or HAIC alone treatment to disease progression or death. PFS will be categorized into intrahepatic PFS and overall PFS.

SECONDARY OUTCOMES:
Treatment efficacy-OS | Through study completion, an average of 1 year
  OS is defined as the time from the date of the first DEB-TACE combined with HAIC or HAIC alone treatment to death
Treatment efficacy-ORR | 6-8 weeks after each treatment
  ORR=CR+PR
Treatment efficacy-DCR | 6-8 weeks after each treatment
  DCR=CR+PR+SD
treatment safety | within 30 days after each treatment
  the frequency of adverse events after treatment

CONTACTS AND LOCATIONS:
Overall Officials: XU zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute